CLINICAL TRIAL: NCT05294016
Title: Smart Bra for Diagnosing Breast Cancer: Pilot Study - CBRA
Brief Title: Smart Bra for Diagnosing Breast Cancer
Acronym: CBRA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Nord Franche-Comte (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2021-04
Record Dates: First submitted 2022-03-15; First posted 2022-03-24 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Breast Cancer; Medical Device
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patient group (Other)
  Interventions: Device: BRA CONNECT device
- Control group (Other)
  Interventions: Device: BRA CONNECT device

INTERVENTIONS:
Device: BRA CONNECT device — skin thermal analysis for the detection of breast abnormalities

SUMMARY:
This project aims to assess the ability of a portable and connected medical device to detect breast abnormalities, for breast cancer screening. It will accelerate technological progress in the face of breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Non-specific invasive carcinoma diagnosed by biopsy
* X-ray images available
* Tumor larger than 1 cm assessed radiologically and/or by ultrasound and/or clinically
* Patient with a breast size compatible with the study bra size

Exclusion Criteria:

* Contralateral breast cancer
* Inflammatory breast cancer
* History of cosmetic or plastic surgery (mastopexy, prosthesis, lipomodelling)
* History of breast cancer or mastectomy
* Presence of dermatological pathology or breast skin ulceration
* Hematoma post biopsy
* History of thoraco-abdominal radiotherapy
* Known allergy to one of the materials of the device
* Fever (body temperature > 37.8°C)
* Pacemaker port

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-04-13 (Actual); Primary Completion 2025-10-28 (Estimated); Study Completion 2025-11-28 (Estimated)

PRIMARY OUTCOMES:
Assess the ability of the device to detect breast abnormalities or not, in healthy women or women with a non-specific invasive carcinoma diagnosed. | 20 minutes of recording
  Sensitivity and specificity of the device to detect a breast abnormality

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - ICANS (Institut de Cancérologie de Strasbourg), Strasbourg
  - Hôpital Nord Franche-Comté, Trévenans

IPD SHARING:
Plan to Share IPD: No